CLINICAL TRIAL: NCT02495935
Title: Feasibility and Efficacy of Transcorneal Electrical Stimulation (TES) for the Treatment of Amblyopia
Brief Title: Transcorneal Electrical Stimulation (TES) for the Treatment of Amblyopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wills Eye (Other)
Collaborators: Harold P. Koller, MD (Unknown); Judith B. Lavrich, MD (Unknown)
Responsible Party: Principal Investigator, Dr. Leonard B. Nelson, MD, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#15-478
Record Dates: First submitted 2015-07-06; First posted 2015-07-13 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Amblyopia
Keywords: TES; Transcorneal Electrical Stimulation; Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- OkuStim® (Experimental): The OkuStim® group will undergo 30-minute treatments once a week for 12 weeks at 200% threshold level according to their individual phosphene threshold (IPT) readings from the OkuStim® device at the pre-treatment visit (week 1). Rectangular biphasic current pulses (1-ms positive, directly followed by 1-ms negative) will be applied at a frequency of 20 Hz.
  Interventions: Device: OkuStim®
- Sham-OkuStim® (Sham Comparator): Subjects in the Sham-OkuStim® group will wear treatment glasses and corneal electrodes for 30 minutes weekly for 12 weeks, but corneal electrodes will not be activated.
  Interventions: Device: Sham-OkuStim®

INTERVENTIONS:
Device: OkuStim® — Transcorneal Electrical Stimulation delivered by the Okuvision Stimulation Set manufactured by Okuvision GmbH, Reutlingen, Germany
  Other Names: TES; Transcorneal Electrical Stimulation
  Arms: OkuStim®
Device: Sham-OkuStim® — Transcorneal Electrical Stimulation delivered by the Okuvision Stimulation Set manufactured by Okuvision GmbH, Reutlingen, Germany
  Arms: Sham-OkuStim®

SUMMARY:
This is a prospective, randomized, parallel group sham-controlled blinded clinical trial to assess the feasibility and efficacy of transcorneal electrical stimulation (TES) in the improvement of visual function outcomes in adults with amblyopia. The trial will assess the treatment effect of TES to Sham TES in the amblyopic eye of affected patients.

DETAILED DESCRIPTION:
Amblyopia is defined as a decrease in visual acuity in one eye, despite the correction of any refractive error with glasses and in the absence of any ophthalmoscopically visible lesion of the retina, especially of the macular region. Amblyopia is associated with histologic and electrophysiologic abnormalities in the visual pathways.

Transcorneal electrical stimulation (TES), through neural stimulation, works by non-invasively stimulating the retina via passage of electrical current directly to the retina, bypassing the usual light activation pathway, resulting in the activation of the same areas of the brain as would be activated with a light stimulus alone. Electrical stimulation with TES has shown potential in recent reports as an efficacious treatment modality to improve visual function.

The success of electrical stimulation in neurodegenerative disorders provides a reasonable rationale and significant precedent to investigate its potential for use in disorders of the visual processing system, which functions via an integration of biochemical and electrical interactions transmitted from the retina.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosis of amblyopia made by the principal investigators.
3. Best corrected visual acuity in the amblyopic eye equal to or worse than 20/70
4. Willing and able to give informed consent and to participate for the full duration of the study.
5. Strabismus less than 10 prism diopters.

Exclusion Criteria:

1. Any other significant ophthalmologic disorder or condition with relevant effect upon visual function as evaluated by principal investigator. (eg. Retinal degeneration, proliferative diabetic retinopathy, age related macular degeneration, optic nerve abnormality)
2. Women who are pregnant or women with childbearing potential who are unwilling to use medically acceptable means of birth control for study duration.
3. Presence of a pacemaker, any metal artifacts in head and trunk, any history of epileptic seizure or severe psychiatric disease (schizophrenia, etc.)
4. Inability to detect phosphenes above 0.5mA at time of threshold detection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Mean change in Best Corrected Visual Acuity (ETDRS letters) | 16 weeks
  Change From Baseline in Best Corrected Visual Acuity (BCVA) as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) to Week 16 (4 weeks post last treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- WillsEye Hospital, Philadelphia, Pennsylvania, United States